CLINICAL TRIAL: NCT07313917
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase Ⅱ Clinical Trial to Evaluate the Efficacy and Safety of LP-003 Injection in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: A Study to Evaluate the Efficacy and Safety of LP-003 Injection in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P10-LP003-12
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LP-003 300 mg group (Experimental): Participants will receive subcutaneous injection of LP-003 Injection at a dose of 300 mg once every 12 weeks.
  Interventions: Biological: LP-003 Injection
- LP-003 450 mg group (Experimental): Participants will receive subcutaneous injection of LP-003 Injection at a dose of 450 mg once every 12 weeks.
  Interventions: Biological: LP-003 Injection
- Placebo (Placebo Comparator): Participants will receive subcutaneous injection of placebo Injection once every 12 weeks.
  Interventions: Biological: Placebo of LP-003

INTERVENTIONS:
Biological: LP-003 Injection — s.c. injection, Q12W
  Arms: LP-003 300 mg group; LP-003 450 mg group
Biological: Placebo of LP-003 — s.c. injection, Q12W
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase II clinical trial. Its primary objective is to explore and preliminarily evaluate the efficacy and safety of LP-003 Injection in the treatment of participants with chronic rhinosinusitis with nasal polyps (CRSwNP), as well as to investigate its pharmacokinetic (PK), pharmacodynamic (PD) profiles, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the study and voluntarily signing the Informed Consent Form (ICF);
2. Aged 18 to 75 years (inclusive) at the time of signing the ICF, regardless of gender;
3. Diagnosis of bilateral chronic rhinosinusitis with nasal polyps (CRSwNP);
4. Persistence of the following symptoms for ≥ 4 weeks prior to the screening/run-in period:

   * Nasal congestion;
   * Any one of the other symptoms: mucoid or mucopurulent nasal discharge, head and facial distension/pain, hyposmia or anosmia;
5. Nasal Polyp Score (NPS) ≥ 5 points, with each nasal cavity scoring at least ≥ 2 points during the screening/run-in period and prior to randomization;
6. Participants report moderate to severe nasal congestion during the screening/run-in period and prior to randomization:

   * Nasal Congestion Score (NCS) of 2 or 3 points at the screening/run-in period (Visit 1, V1);
   * Mean weekly NCS ≥ 2 points prior to randomization;
7. With bilateral CRSwNP despite prior treatment with systemic corticosteroids (SCS) such as oral corticosteroids (OCS) within 2 years prior to screening; and/or has contraindications to SCS treatment or is intolerant to SCS; and/or has undergone nasal polypectomy within 6 months prior to screening, with persistent bilateral CRSwNP.
8. Has been on a stable dosage of intranasal corticosteroids (INCS) for at least 4 weeks prior to screening;
9. Demonstrates ≥80% adherence to mometasone furoate nasal spray (MFNS) administration during the run-in period (with a minimum of 14 days of use).

Exclusion Criteria:

1. Concurrent other nasal diseases or nasal symptoms;
2. Acute upper respiratory tract infection at screening, which the investigator assesses may affect nasal symptom scoring;
3. Severe infection requiring intravenous antibiotics and/or hospitalization within 4 weeks prior to randomization that has not yet resolved, or active infection requiring oral antibiotics within 2 weeks prior to randomization that has not yet resolved; the investigator assesses that enrollment of the participant may pose uncontrollable risks;
4. Concurrent active parasitic infection (e.g., helminths) or suspected parasitic infection;
5. Known or suspected history of immunosuppression, including a history of invasive opportunistic infections (e.g., histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis); or participants with a history of such infections that have resolved but are assessed by the investigator as likely to recur frequently;
6. Any severe or unstable disease that the investigator believes may affect the participant's safety during the study and/or hinder the participant from completing the study;
7. Has any severe or unstable disease that, in the investigator's judgment, may affect the safety of the trial participant during the study and/or preclude the participant from completing the study, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, autoimmune, hematological, or psychiatric disorders.
8. Current or prior receipt of the following treatments:

   * Use of traditional Chinese medicine (TCM) or proprietary Chinese medicines for chronic rhinosinusitis within 1 week prior to screening;
   * Use of medium- or short-acting systemic corticosteroids (SCS) within 4 weeks prior to randomization, or long-acting SCS within 6 weeks prior to randomization;
   * Receipt of any systemic monoclonal antibody therapy [e.g., Stapokibart, Dupilumab, Mepolizumab, Omalizumab, Tezepelumab, etc.] within 10 weeks prior to randomization or within 5 half-lives (whichever is longer);
   * Use of systemic immunosuppressants within 4 weeks prior to randomization or within 5 half-lives (whichever is longer);
   * Initiation of leukotriene receptor antagonist (LTRA) therapy within 4 weeks prior to randomization (participants who have been receiving stable-dose LTRA therapy for at least 4 weeks prior to randomization are eligible for enrollment);
9. For participants with concurrent asthma, the forced expiratory volume in 1 second (FEV1) as a percentage of predicted value ≤ 50% during the screening/run-in period;
10. Known allergy or intolerance to any component of the investigational product and/or mometasone furoate nasal spray;
11. Pregnant or lactating females;
12. Any other conditions that the investigator deems inappropriate for the participant to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Nasal Polyps Score (NPS) at Week 24 | Week 24
  NPS is a bilateral endoscopic assessment scale for nasal polyposis, where each nasal cavity is scored from 0 to 4. The total score is the sum of the left and right sides, ranging from 0 to 8, with higher scores indicating more severe nasal polyp disease.
Change from baseline in Nasal Congestion Score (NCS) at Week 24 | Week 24
  The NCS is a patient-reported outcome measure using a 0-3 point Verbal Rating Scale (VRS). Patients rate their nasal congestion severity as 0 (no symptoms), 1 (mild symptoms), 2 (moderate symptoms), or 3 (severe symptoms). The total score ranges from 0 to 3, with higher scores indicating more severe nasal congestion.

SECONDARY OUTCOMES:
Change from baseline in NPS at each assessment visit (excluding Week 24) | Up to approximately 56 weeks
Percentage of participants with a ≥1-point improvement in NPS from baseline | Up to approximately 56 weeks
Percentage of participants with a ≥2-point improvement in NPS from baseline | Up to approximately 56 weeks
Change from baseline in NCS at each assessment visit (excluding Week 24) | Up to approximately 56 weeks
Percentage of participants with a ≥1-point improvement in NCS from baseline | Up to approximately 56 weeks
Change from baseline in Total Score of 22-Items Sinonasal Outcome Test (SNOT-22) | Up to approximately 56 weeks
  The SNOT-22 is a validated 22-items questionnaire to assess the impact of chronic rhinosinusitis on health-related quality of life (HRQoL) with a recall period of 2 weeks. There are 5 domains that could be described within SNOT-22, including nasal, ear, sleep, general and practical, and emotional; each domain was scored on a 6-category scale which ranged from 0: no problem to 5: problem as bad as it can be. The total score was the sum of response to each of the 22 questions and ranged from 0 (no disease) to 110 (worst disease), higher scores indicated worse HRQoL.
Incidence of adverse events (AEs) | Up to approximately 56 weeks
Number of patients with anti-drug antibodies (ADA) | Up to approximately 56 weeks
Serum concentrations of LP-003 | Up to approximately 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, China